CLINICAL TRIAL: NCT06608615
Title: Investigation of the Instant Effect of Rigid and Kinesio Taping Techniques on Physical Performance, Gait and Physiological Expenditure Index in Stroke Individuals With Foot Drop
Brief Title: the Instant Effect of Rigid and Kinesio Taping Techniques in Stroke Individuals With Foot Drop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Saniye Aydoğan Arslan, Kırıkkale University, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KırıkkaleüniylÖmerKaya; Ömer Kaya (Other: Kırıkkale Üniversitesi)
Record Dates: First submitted 2024-05-29; First posted 2024-09-23 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Physical Performance, Gait and Physiological Expenditure Index in Stroke Patients
Keywords: Rigid Taping; Kinesio Taping; Drop Foot Gait; Stroke
MeSH Terms: conditions — Gait Disorders, Neurologic; Stroke | interventions — Functional Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping Group (Experimental): Persons who will undergo kinesio taping
  Interventions: Other: Kinesio Taping
- Rigid Taping group (Experimental): Persons to whom rigid taping will be performed
  Interventions: Other: Rigid Taping

INTERVENTIONS:
Other: Kinesio Taping — Facilitation (Functional) Technique for Tibialis Anterior Muscle: The patient sits with his leg extended. The ankle is placed in eversion and dorsi flexion. After one end of the I tape is adhered to the upper part of the Tibia, the other end is adhered to the dorsal surface of the foot with almost 100% tension. During the application, origin and insertion points are considered as the beginning and end. Then, plantar fexion is performed on the ankle and the remaining non-stick part is glued.
  Functional Correction Technique: Correction technique is used to ensure full contact of the foot with the ground. The subtalar joint is positioned in eversion and taping is applied starting from under the medial malleolus, without tension until the lateral outer edge of the calceneus, and then with 100% tension, continuing until 10-15 cm below the head of the fibula. No tension is applied in the last 5 cm
  Other Names: Functional Correction Technique; Facilitation (Functional) Technique for Tibialis Anterior Muscle
  Arms: Kinesio Taping Group
Other: Rigid Taping — Talus Stabilization Taping: The affected ankle of the person to be taped was placed on a chair and asked to bring this foot to a neutral position by advancing the tibia over the foot through knee flexion while standing. Starting from the talus of the ankle, maximum tension was applied towards the medial and lateral malleolus.
  Inversion Lock: This lock looks like an inverted 6 when viewed from the front and is used to restrict inversion movement. After the underwrap and anchor were applied, the tape was applied starting from the outer malleolus level. It was glued on itself by proceeding diagonally in front of the foot, passing it in front of the inner malleolus, passing under the foot and in front of the outer malleolus and closing the subtalar area, and the taping was completed by making an anchor on the upper side.
  Other Names: Talus Stabilization Taping; Inversion Lock
  Arms: Rigid Taping group

SUMMARY:
Stroke individuals with foot drop experience poor physical performance and walking problems. Physiological energy consumption also increases due to balance and walking problems. The aim of this study is to investigate the immediate effects of rigid and kinesio taping techniques on physical performance, gait and physiological expenditure index in stroke individuals with foot drop, and also to examine whether these approaches are superior to each other.

As a result of this study, it was seen that Rigid Taping and Kinesio Taping were effective in stroke individuals with foot drop. When we compared the groups, it was determined that both taping methods produced similar effects.

DETAILED DESCRIPTION:
Stroke individuals with foot drop experience poor physical performance and walking problems. Physiological energy consumption also increases due to balance and walking problems. The aim of this study is to investigate the immediate effects of rigid and kinesio taping techniques on physical performance, gait and physiological expenditure index in stroke individuals with foot drop, and also to examine whether these approaches are superior to each other.

40 individuals diagnosed with hemorrhagic or ischemic stroke were included in the study. Individuals were divided into two groups: Rigid Taping Group (n=20) and Kinesio Taping Group (n=20). The physical performances of the individuals participating in the study were evaluated with the One-Leg Standing Test, Timed Up and Go Test (TUG) and the Sit-Up-from-Chair Test (SUCT), their walking speed was evaluated with the 10 Meter Walk Test, and the spatiotemporal characteristics of the gait were evaluated with gait analysis on powdered ground. Physiological Expenditure Index (FHI) was calculated with 6 Minute Walk Test (6MWT) results. Evaluations were recorded by the same physiotherapist before and after taping.

As a result of this study, it was seen that Rigid Taping and Kinesio Taping were effective in stroke individuals with foot drop. When we compared the groups, it was determined that both taping methods produced similar effects. We believe that adding rigid or kinesio taping applications for foot drop to the rehabilitation program of stroke individuals with drop foot will increase the success of the treatment.

ELIGIBILITY:
Being diagnosed with ischemic or hemorrhagic stroke, Not having cooperation and communication problems, Stroke individuals with foot drop and those with a MAS score of 2 or less, Those who score 0-3 on the Modified Rankin Scale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Timed up and go test | 3 minutes
  "The timed up and go measures, in seconds, the time taken by an individual to stand up from a standard arm chair (approximate seat height of 46 cm), walk a distance of 3 metres, turn, walk back to the chair and sit down again. The subject wears his regular footwear and uses his customary walking aid (none, cane, or walker). No physical assistance is given. He starts with his back against the chair, his arms resting on the chair's arms and his walking aid at hand. He is instructed that, on the word "go", he is to get up and walk at a comfortable and safe pace to a line on the floor 3 metres away, turn, return to the chair and sit down again. The subject walks through the test once before being timed in order to become familiar with the test.both taping methods produced similar effects.
10 metre walking test | 1 minutes
  Gait speed was based on the average of two trials of the 10-m TWT in order to reduce measurement error. Patients were instructed to walk independently from other people as fast and safely as possible, and were allowed to use a walking aid if needed. The 10 metres had to be free of obstacles and turns. program of stroke individuals with drop foot will increase the success of the treatment.
Sit up and chair test | 1 minutes
  ubjects began the test sitting on a 47 cm-high chair, positioned with the feet hip width apart, toes under knees and arms folded across their chest. The investigators recorded the length of time to the nearest tenth of a second it took for subjects to rise and sit back down five consecutive times without the use of their arms. Participants were given one practice trial to familiarize themselves with the procedure.kullanımında etkili olduğunu göstermektedir.
six minute walk test | 10 minutes
  The functional capacity of the individuals was evaluated with 6MWT. The measurements were made in line with the recommendations of the American Thoracic Society. The individuals were asked to walk in a 30-m corridor at their own walking speed for 6 min as far as possible. The individuals were allowed to stop and rest during the test, which was repeated twice every other day. The maximum 6 min walking dis- tance was recorded in meters.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)